CLINICAL TRIAL: NCT00604370
Title: VTE Prophylaxis Across the Continuum of Care: High Risk Patients at Hospital Discharge
Brief Title: Retrospective Study to Review Patients at Risk for VTE at Hospital Discharge
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Samuel Z.Goldhaber, MD, Director, VTE Research Group, Brigham and Women's Hospital
Other Study IDs: 2006-P-001981
Record Dates: First submitted 2007-12-28; First posted 2008-01-30 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Acutely ill medical and surgical patients who were hospitalized at BWH, and at-risk for VTE, but were not treated with prophylaxis at hospital discharge.
- 2: Acutely ill medical and surgical patients who were at risk for VTE at time of hospital discharge and prescribed a prophylaxis strategy.

SUMMARY:
An investigator initiated study exploring VTE prophylaxis at the time of hospital discharge.

DETAILED DESCRIPTION:
It appears likely that many patients will remain at risk for VTE at the time of hospital discharge. These risks will go unrecognized, and discharge prophylaxis orders will not be prescribed.

To test this hypothesis, we will perform a retrospective review of approximately 2,500 patients at Brigham and Women's Hospital at risk for VTE at the time of hospital discharge to determine what proportion received VTE prophylaxis. We will correlate the implementation of discharge VTE prophylaxis with the occurrence of symptomatic DVT and pulmonary embolism within 90 days of hospital discharge.

We will also conduct a substudy of this patient population to determine adherence to VTE prophylaxis among hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Acutely ill medical and surgical patients with a risk score of 4 or greater without prophylaxis or a risk score of 4 or greater with anticoagulation at hospital discharge.

Exclusion Criteria:

* None.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acutely ill medical and surgical patients who were hospitalized at BWH and who are at risk for DVT.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic PE/DVT within 90 days of hospital discharge. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital